CLINICAL TRIAL: NCT02286453
Title: Clinical Efficacy and Safety of Benjakul Recipe in Treating Primary Osteoarthritis of Knee Compared With Diclofenac (Clinical Trial Phase II)
Brief Title: Clinical Efficacy and Safety of Benjakul Recipe in Treating Primary Osteoarthritis of Knee Compared With Diclofenac
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thammasat University (Other)
Collaborators: Thai Traditional Medical Knowledge Fund (Other Government)
Responsible Party: Principal Investigator, Patamaporn Rachawat, Piya Pinsornsak, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTU-EC-ES-6-152/56; TCTR20140816001 (Registry Identifier: Thai Clinical Trials Registry)
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis of The knee; Benjakul; Alternative Medicine
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Benjakul
  Interventions: Drug: Benjakul recipe
- 2 (Active Comparator): diclofenac
  Interventions: Drug: diclofenac

INTERVENTIONS:
Drug: Benjakul recipe — Benjakul recipe capsule at dose of 100 mg three times a day after meal daily for 28 days
  Arms: 1
Drug: diclofenac — diclofenac capsule at dose of 25 mg three times a day after meal daily for 28 days
  Arms: 2

SUMMARY:
Efficacy and adverse effects of Benjakul recipe in Treating Primary Osteoarthritis of Knee Compared with Diclofenac. This study was designed as double blind, randomized controlled trial. Approval from the ethical committee of Human Research Ethics Committee of Thammasat University (No: 1 Faculty of Medicine)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary osteoarthritis of knee with grade I-III of Kellgren & Lawrence criteria
2. Not during breast feeding
3. Not during pregnancy with a good contraception
4. Volunteer have a normal Complete Blood Count laboratory, lipid profiles,liver function tests and renal funtion tests
5. Do not abuse drugs
6. Good cooperation

Exclusion Criteria:

1. BMI > 32
2. History of peptic ulcer, Gastroesophageal reflux disease (GERD), heart disease, liver disease or kidney disease
3. History of allergy diclofenac or allergy herbal medicine

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pain score | 28 days
  Pain score from Visual analog scale

SECONDARY OUTCOMES:
Pain score | 28 days
  Pain score from Modified WOMAC score (from Modified Thai WOMAC index)

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University (Ruangsit campus), Khlong Luang, Changwat Pathum Thani, Thailand